CLINICAL TRIAL: NCT02637388
Title: The Effect of a Breakfast Meal Containing 4g Oat Beta-glucan on Perceived Satiety and ad Libitum Food Intake in Normal-weight and Overweight Subjects. A Double-blinded, Randomized, Placebo-controlled Cross-over Study.
Brief Title: Effects of Beta-glucan on Energy Intake and Satiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Queen Margaret University (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Suzanne Zaremba, Principle Investigator, Queen Margaret University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: QueenMUsz2
Record Dates: First submitted 2015-12-11; First posted 2015-12-22 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: Appetite; Beta-glucans; Energy Intake; Glucagon-Like Peptide 1; Glucose; Insulin; Incretins
MeSH Terms: conditions — Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Comparator: Control Breakfast (Placebo Comparator): Breakfast cereal and yoghurt only (placebo, negative control)
  Interventions: Dietary Supplement: Control Breakfast
- Experimental: beta-Glucan Breakfast (Experimental): Breakfast cereal and yoghurt with the addition of 4g beta-glucan (14.7g Oatwell28 powder)
  Interventions: Dietary Supplement: Oatwell28 Oatwell Original Powder

INTERVENTIONS:
Dietary Supplement: Oatwell28 Oatwell Original Powder
  Arms: Experimental: beta-Glucan Breakfast
Dietary Supplement: Control Breakfast — Isocaloric breakfast without added beta-glucans
  Arms: Placebo Comparator: Control Breakfast

SUMMARY:
The purpose of this study is to address the effect of consuming 4g of soluble fibre beta-glucan at breakfast on satiety and food intake.

DETAILED DESCRIPTION:
Satiation and satiety are part of the body's complex appetite control system that ultimately play a role in limiting energy intake. Satiation is referred to as the process that leads to the termination of eating, which may be accompanied by feelings of satisfaction. Satiety is the feeling of fullness that persists after eating, with the potential to suppress further energy intake until hunger returns. There is evidence to suggest that increasing gastro-intestinal viscosity improves appetite control and reduces subsequent food intake. Beta-glucan is a soluble fibre proposed to behave this way.

In this double-blinded, randomized, crossover trial, subjective appetite sensations will be measured and blood will be collected at specific time points during the two arms in order to determine hormonal responses. Ad libitum food intake will be recorded. Food diaries will be used to measure dietary intakes.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females, aged 18-50 years
* BMI of 20.0 - 29.9 kg/m2 at screening
* Subjects who usually consume breakfast
* Subject is willing to stick to his/her normal habitual diet, excluding the consumption of any unusual high energy-rich or fat-rich meals or undergo periods of fasting during the study period.
* Subject is willing to abstain from strenuous exercise, consume alcoholic drinks and caffeine containing food/drinks 24hours before study days and during study days.
* Ability to pass the Dutch Eating Behaviour Questionnaire (Van Strein et al. 1986) to measure dietary restraint, disinhibition and hunger
* Subjects understands the study procedures and signs the informed consent to participate in the study
* Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the investigator on the basis of medical history or parameters measured during screening.
* Subject has been stable in body-weight within the last 6 months.
* Female subjects are willing to use a contraceptive method to avoid pregnancy during the study period.

Exclusion Criteria:

* Postmenopausal females
* Smokers
* Individuals who suffer from (or taking medication for) cardiovascular disease or gastrointestinal disease, including hypertension, hypercholesterolemia, hyperlipidaemia, Crohn's Disease, Irritable bowel syndrome, etc.
* Impaired glucose tolerance/Diabetes mellitus (Fasting blood glucose of ≥5.6mmol/l or 100mg/dL as per NHS criteria)
* Haemoglobin measurements of <120g/L for females and <130g/L for males (as per WHO criteria for anaemia)
* Pregnancy or breastfeeding
* Those who consume a high fibre diet - consumption of more than 20g/day - Individuals who have known food allergies to ingredients used in study meals (wheat, cow's milk, ham, dairy)
* Needle phobia
* Subjects who are on hypocaloric/hypercaloric diet aiming for weight loss/gain.
* Recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >60g (men) / 40g (women) pure alcohol per day (1.5 l / 1 l beer resp. 0.75 l / 0.5 l wine).
* Subject has donated more than 300 mL of blood during the three months prior to screening.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Variation in energy intakes | 1 day
  Ad libitum food intake (kilocalories) will be determined during an 'all you can' eat buffet lunch. Food intakes will be measured over 5 days; 3 days prior to the study day, on the day of the study and the day after.

SECONDARY OUTCOMES:
Variation in the feelings of appetite | -30, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150 minutes
  Measure of the satiating effect for each breakfast with Visual Analog Scale (Area Under the Curve) over time for subjective appetite parameters
Variation in GLP-1 | 0, 30, 60, 90 minutes
  Measure plasma total glucagon-like peptide 1 (GLP-1) area under the curve (AUC) over time.
Variation in insulin | 0, 30, 60, 90 minutes
  Measure plasma insulin (pg/mL) area under the curve (AUC) over time.
Variation in glucose | 0, 30, 60, 90, 120 minutes
  Measure blood glucose (mmol/L) area under the curve (AUC) over time.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Zaremba, Principal Investigator — Queen Margaret University
Locations (1):
- Queen Margaret University, Edinburgh, Musselburgh, East Lothain, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barone Lumaga R, Azzali D, Fogliano V, Scalfi L, Vitaglione P. Sugar and dietary fibre composition influence, by different hormonal response, the satiating capacity of a fruit-based and a beta-glucan-enriched beverage. Food Funct. 2012 Jan;3(1):67-75. doi: 10.1039/c1fo10065c. Epub 2011 Nov 4. PMID 22057424
- [Background] Vitaglione P, Lumaga RB, Montagnese C, Messia MC, Marconi E, Scalfi L. Satiating effect of a barley beta-glucan-enriched snack. J Am Coll Nutr. 2010 Apr;29(2):113-21. doi: 10.1080/07315724.2010.10719824. PMID 20679146
- [Background] Vitaglione P, Lumaga RB, Stanzione A, Scalfi L, Fogliano V. beta-Glucan-enriched bread reduces energy intake and modifies plasma ghrelin and peptide YY concentrations in the short term. Appetite. 2009 Dec;53(3):338-44. doi: 10.1016/j.appet.2009.07.013. Epub 2009 Jul 23. PMID 19631705
- [Background] Juvonen KR, Salmenkallio-Marttila M, Lyly M, Liukkonen KH, Lahteenmaki L, Laaksonen DE, Uusitupa MI, Herzig KH, Poutanen KS, Karhunen LJ. Semisolid meal enriched in oat bran decreases plasma glucose and insulin levels, but does not change gastrointestinal peptide responses or short-term appetite in healthy subjects. Nutr Metab Cardiovasc Dis. 2011 Sep;21(9):748-56. doi: 10.1016/j.numecd.2010.02.002. Epub 2010 Jun 4. PMID 20605427
- [Background] Huang XF, Yu Y, Beck EJ, South T, Li Y, Batterham MJ, Tapsell LC, Chen J. Diet high in oat beta-glucan activates the gut-hypothalamic (PYY(3)(-)(3)(6)-NPY) axis and increases satiety in diet-induced obesity in mice. Mol Nutr Food Res. 2011 Jul;55(7):1118-21. doi: 10.1002/mnfr.201100095. Epub 2011 Jun 20. PMID 21688388
- [Background] Steinert RE, Beglinger C, Langhans W. Intestinal GLP-1 and satiation: from man to rodents and back. Int J Obes (Lond). 2016 Feb;40(2):198-205. doi: 10.1038/ijo.2015.172. Epub 2015 Aug 28. PMID 26315842
- [Background] Steinert RE, Schirra J, Meyer-Gerspach AC, Kienle P, Fischer H, Schulte F, Goeke B, Beglinger C. Effect of glucagon-like peptide-1 receptor antagonism on appetite and food intake in healthy men. Am J Clin Nutr. 2014 Aug;100(2):514-23. doi: 10.3945/ajcn.114.083246. Epub 2014 Jun 25. PMID 24965303